CLINICAL TRIAL: NCT00663234
Title: Phase I/II Safety and Efficacy Investigation of Atorvastatin for Treatment of PI-Associated Increased LDL Cholesterol in HIV-Infected Children and Adolescents
Brief Title: IMPAACT P1063: Safety and Effectiveness of Atorvastatin in HIV Infected Children and Adolescents With Hyperlipidemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to administrative reasons.
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT P1063; U01AI068632 (NIH); 10167
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections; Hyperlipidemia
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Age 10 to 14 (Experimental): Participants ages 10 to 14 years receiving oral atorvastatin for 48 weeks while on a stable antiretroviral regimen
  Interventions: Drug: Atorvastatin
- Age 15 to 23 (Experimental): Participants ages 15 to 23 years receiving oral atorvastatin for 48 weeks while on a stable antiretroviral regimen
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 10 mg to 20 mg atorvastatin taken orally once daily. Dosage is dependent on efficacy criteria.
  Other Names: Lipitor

SUMMARY:
Treatment of HIV with combination antiretroviral regimens frequently results in the suppression of HIV viral load, significant immune recovery, and delayed disease progression. However, treatment with these regimens, particularly protease inhibitors (PIs), has been associated with significant increases in cholesterol and triglycerides in HIV-infected adults and children. The purpose of this study was to evaluate the safety and effectiveness of escalating doses of atorvastatin, a FDA-approved drug which lowers cholesterol and triglyceride levels, in HIV-infected children receiving stable antiretroviral regimens.

DETAILED DESCRIPTION:
Antiretroviral regimens, particularly those containing PIs, often cause hyperlipidemia, which is an increase in the amount of fat (such as cholesterol and triglycerides) in the blood. These increases can lead to heart disease and pancreatitis. Although the mechanism by which PIs cause hyperlipidemia is not clearly understood, there are medications to combat this side effect. The primary purpose of this study was to evaluate the safety and effectiveness of escalating doses of atorvastatin, based on low-density lipoprotein cholesterol (LDL-C) levels, in HIV-infected children receiving stable antiretroviral therapy.

Participants were assigned to one of two groups based on age (10 to 14 years or 15 to 23 years) and were treated for a maximum of 48 weeks. The first six participants enrolled in the study were in the 15 to 23 year old age group. Once safety data through week 8 on these 6 participants was analyzed, the remaining participants were enrolled. All participants received atorvastatin in combination with a stable antiretroviral regimen. Each participant was followed independently according to a dose escalation algorithm for atorvastatin. Participants began dosing at 10 mg daily. If efficacy criteria were not met, dosing increased to 20 mg daily at week 8. Since dose escalations were done within subject, safety and efficacy rates were presented for the dose-escalation strategy overall and not for individual doses. Atorvastatin was provided by the study, but antiretrovirals were not.

Study visits occurred at study entry and weeks 4, 8, 12, 24, 36, and 48. Safety labs were collected at all study visits. Blood collection for lipid measurements occurred at weeks 4, 12, 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of HIV-1 infection
* CD4 % of at least 15 at screening
* HIV-1 viral load of less than 10,000 copies/ml at screening
* On a stable antiretroviral therapy regimen for at least 6 months
* Tanner stage of 2 or higher
* At least two LDL-C measurements of 130 mg/dL or higher over the 6 months prior to screening and after documented attempts at modifying diet and other risk factors. More information on this criterion can be found in the protocol.
* Able to fast overnight for 8 hours
* Negative pregnancy test at screening
* Agree to use two appropriate forms of contraception (female participants). More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Certain abnormal laboratory values
* Any laboratory or unresolved clinical toxicity of Grade 3 or higher
* Unlikely to remain on current antiretroviral therapy for at least six months after study entry
* Use of statin, fibrate, or niacin within 3 months prior to study entry
* Evidence of chronic ongoing myositis or history of myopathy or neuromuscular disorder
* Symptomatic peripheral neuropathy within 6 months prior to study entry
* Pharmacologic treatment for depression or other mental disorder excluding Attention Deficit Disorder within 30 days prior to study entry
* Presence of an active CDC Stage C opportunistic infection or serious bacterial infection requiring therapy within 2 weeks prior to screening.
* Chemotherapy for malignancy within 3 months prior to study entry
* Hepatitis B Surface Antigen positive
* Hepatitis C viremia
* Insulin-dependent diabetes mellitus
* Required treatment with an agent contraindicated with either atorvastatin or PIs. More information on this criterion can be found in the protocol.
* Pregnant or breastfeeding

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Melvin, MD, Study Chair — Seattle Children's Hospital; Marilyn Crain, MD, MPH, Study Chair — University of Alabama at Birmingham
Locations (11):
- United States (11):
  - Univ. of Colorado Denver NICHD CRS (5052), Aurora, Colorado
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS (4201), Miami, Florida
  - University of South Florida Tampa (5018), Tampa, Florida
  - Chicago Children's CRS (4001), Chicago, Illinois
  - Tulane University (5095), New Orleans, Louisiana
  - Boston Medical Center Ped. HIV Program NICHD CRS (5011), Boston, Massachusetts
  - New York University NY (5012), New York, New York
  - Metropolitan Hospital (5003), New York, New York
  - Bronx-Lebanon Hospital IMPAACT CRS (6901), The Bronx, New York
  - St. Jude/UTHSC CRS (6501), Memphis, Tennessee
  - Texas Children's Hosp. CRS (3801), Houston, Texas

REFERENCES:
- [Background] Kamin D, Hadigan C. Hyperlipidemia in children with HIV infection: an emerging problem. Expert Rev Cardiovasc Ther. 2003 May;1(1):143-50. doi: 10.1586/14779072.1.1.143. PMID 15030304
- [Background] Penzak SR, Chuck SK. Management of protease inhibitor-associated hyperlipidemia. Am J Cardiovasc Drugs. 2002;2(2):91-106. doi: 10.2165/00129784-200202020-00003. PMID 14727985
- [Background] Solorzano Santos F, Gochicoa Rangel LG, Palacios Saucedo G, Vazquez Rosales G, Miranda Novales MG. Hypertriglyceridemia and hypercholesterolemia in human immunodeficiency virus-1-infected children treated with protease inhibitors. Arch Med Res. 2006 Jan;37(1):129-32. doi: 10.1016/j.arcmed.2005.05.013. PMID 16314198
- [Background] The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between August 31, 2009 (date first participant enrolled) and December 16, 2013 (date last participant enrolled).
Groups:
- Atorvastatin: 10 mg to 20 mg atorvastatin taken orally once daily. Dosage starts at 10 mg and is increased to 20 mg at week 8 if efficacy criteria is not met at week 4.
Period: Overall Study
Arm/Group | Atorvastatin
Started | 28
Dose Increased to 20 mg at Week 8 | 10
Completed | 27
Not Completed | 1
Not completed — Not willing to adhere to requirements | 1

BASELINE CHARACTERISTICS:
Population: All participants who initiated Atorvastatin were included in the baseline characteristics.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (4)
Age, Customized [Number; unit: participants]
  10 - <15 years old | 7
  15 - <19 years old | 12
  19 - <24 years old | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 9
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 4
  Black Non-Hispanic | 18
  Hispanic (Regardless of Race) | 5
  Asian, Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 28
CD4 Percent at screening, Categorical [Number; unit: participants]
  15% to <25% | 2
  >=25% | 26
HIV-1 RNA, Categorical [Number; unit: participants]
  >=Lower limit of quantification of assay | 8
  <Lower limit of quantification of assay | 20
Antiretroviral (ARV) Regimen at entry, Categorical [Number; unit: participants] — ARV regimens are categorized based on whether or not they contain Protease Inhibitors (PIs) and/or Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs).
  participants
    At least one PI and at least one NNRTI | 5
    At least one PI and no NNRTI | 17
    At least one NNRTI and no PI | 4
    Other ARV regimen | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Treatment-related Adverse Event (AE)
Description: AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (see references in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening, Grade 5=Death. Relationship to study treatment was determined by the core study team. The primary outcome measure includes any AE of grade 3 or higher and liver function tests (LFTs) of grade 2 or higher.
Time Frame: Study entry to weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 28
percentage of participants
  Week 12 | 3.6 [0.2 to 15.9]
  Week 24 | 3.6 [0.2 to 15.9]
  Week 48 | 7.1 [1.3 to 20.8]

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE)
Description: AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (see references in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening, Grade 5=Death. The primary outcome measure includes any AE of grade 3 or higher and liver function tests (LFTs) of grade 2 or higher.
Time Frame: Study entry to weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 28
percentage of participants
  Week 12 | 21.4 [9.8 to 38.0]
  Week 24 | 21.4 [9.8 to 38.0]
  Week 48 | 28.6 [15.1 to 45.7]

3. Primary Outcome: Percentage of Participants Who Met the LDL Cholesterol (LDL-C) Efficacy Criteria (Intention to Treat)
Description: Efficacy was defined as having LDL-C of 110 mg/dL or less or at least 30% decline in LDL-C from baseline to the specified week.
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated Atorvastatin. If a participant was missing data at a given week, treatment was assumed to be non-efficacious at that week.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 28
percentage of participants
  Week 4 | 60.7 [43.5 to 76.2]
  Week 12 | 46.4 [30.1 to 63.4]
  Week 24 | 57.1 [40.0 to 73.1]
  Week 48 | 53.6 [36.6 to 69.9]

4. Primary Outcome: Percentage of Participants Who Met the LDL Cholesterol (LDL-C) Efficacy Criteria (Data Available)
Description: as for outcome 3
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated study treatment and have LDL-C data available at study entry and the specified week.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 27
percentage of participants
  Week 4 (N=27) | 63.0 [45.3 to 78.3]
  Week 12 (N=27) | 48.2 [31.3 to 65.3]
  Week 24 (N=26) | 61.5 [43.6 to 77.4]
  Week 48 (N=26) | 57.7 [39.8 to 74.2]

5. Primary Outcome: Percentage of Participants Who Met the LDL Cholesterol (LDL-C) Efficacy Criteria (Per Protocol)
Description: as for outcome 3
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who completed the study per protocol (initiated study drug, had LDL-C data available at all required study visits, attended study visits within the protocol-specified window, were dose-escalated according to protocol, and reported adherence to study drug at all study visits).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 13
percentage of participants
  Week 4 | 69.2 [42.7 to 88.7]
  Week 12 | 69.2 [42.7 to 88.7]
  Week 24 | 84.6 [59.0 to 97.2]
  Week 48 | 53.9 [28.7 to 77.6]

6. Primary Outcome: Percentage of Participants Who Met the LDL Cholesterol (LDL-C) Efficacy Criteria and Did Not Experience a Primary Safety Endpoint Attributable to Study Drug
Description: as for outcome 3
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated Atorvastatin and did not experience a primary safety event attributable to Atorvastatin.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 26
percentage of participants
  Week 4 | 57.7 [39.8 to 74.2]
  Week 12 | 50.0 [32.7 to 67.3]
  Week 24 | 57.7 [39.8 to 74.2]
  Week 48 | 53.9 [36.2 to 70.8]

7. Primary Outcome: Percentage of Participants Who Met the LDL Cholesterol (LDL-C) Efficacy Criteria by Age Group
Description: as for outcome 3
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- 10 to 14 Years Old: Participants ages 10 to 14 years receiving oral atorvastatin for 48 weeks while on a stable antiretroviral regimen
  Atorvastatin: 10 mg to 20 mg atorvastatin taken orally once daily. Dosage is dependent on efficacy criteria.
- 15 to 23 Years Old: Participants ages 15 to 23 years receiving oral atorvastatin for 48 weeks while on a stable antiretroviral regimen
  Atorvastatin: 10 mg to 20 mg atorvastatin taken orally once daily. Dosage is dependent on efficacy criteria.
Arm/Group | 10 to 14 Years Old | 15 to 23 Years Old
Number analyzed (Participants) | 7 | 21
percentage of participants
  Week 4 | 71.4 [34.1 to 94.7] | 57.1 [37.2 to 75.5]
  Week 12 | 28.6 [5.3 to 65.9] | 52.4 [32.8 to 71.4]
  Week 24 | 71.4 [34.1 to 94.7] | 52.4 [32.8 to 71.4]
  Week 48 | 71.4 [34.1 to 94.7] | 47.6 [28.6 to 67.2]

8. Primary Outcome: Percentage of Participants Who Met the LDL Cholesterol (LDL-C) Efficacy Criteria by NNRTI Treatment
Description: as for outcome 3
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- NNRTI-exposed: Participant was on at least one non-nucleoside reverse transcriptase inhibitor (NNRTI) at entry.
- NNRTI-unexposed: Participant was not on at least one non-nucleoside reverse transcriptase inhibitor (NNRTI) at entry.
Arm/Group | NNRTI-exposed | NNRTI-unexposed
Number analyzed (Participants) | 9 | 19
percentage of participants
  Week 4 | 66.7 [34.5 to 90.2] | 57.9 [36.8 to 77.0]
  Week 12 | 55.6 [25.1 to 83.1] | 42.1 [23.0 to 63.2]
  Week 24 | 44.4 [16.9 to 74.9] | 63.2 [41.8 to 81.3]
  Week 48 | 55.6 [25.1 to 83.1] | 52.6 [32.0 to 72.6]

9. Primary Outcome: Percent Change in LDL Cholesterol (LDL-C) From Study Entry
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated Atorvastatin and had LDL-C data available at study entry and the specified week.
Measure: Mean (90% Confidence Interval); unit: percentage of LDL-C at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 27
percentage of LDL-C at study entry
  Percent change in LDL-C at Week 4 (N=27) | -30.3 [-34.6 to -26.1]
  Percent change in LDL-C at Week 12 (N=27) | -26.5 [-32.4 to -20.5]
  Percent change in LDL-C at Week 24 (N=26) | -28.0 [-32.7 to -23.4]
  Percent change in LDL-C at Week 48 (N=26) | -26.4 [-33.1 to -19.7]

10. Secondary Outcome: Percent Change in Fasting Total Cholesterol (TC) From Study Entry
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated Atorvastatin and had total cholesterol data available at study entry and the specified week.
Measure: Mean (90% Confidence Interval); unit: percentage of TC at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 27
percentage of TC at study entry
  Percent change in TC at Week 4 (N=27) | -23.8 [-26.8 to -20.8]
  Percent change in TC at Week 12 (N=27) | -21.1 [-25.1 to -17.1]
  Percent change in TC at Week 24 (N=26) | -22.5 [-26.0 to -19.0]
  Percent change in TC at Week 48 (N=26) | -21.5 [-26.4 to -16.6]

11. Secondary Outcome: Percent Change in Triglycerides (TG) From Study Entry
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated Atorvastatin and had triglycerides data available at study entry and the specified week.
Measure: Mean (90% Confidence Interval); unit: percentage of TG at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 27
percentage of TG at study entry
  Percent change in TG at Week 4 (N=27) | -9.5 [-20.4 to 1.4]
  Percent change in TG at Week 12 (N=27) | -12.6 [-19.5 to -5.7]
  Percent change in TG at Week 24 (N=26) | -11.3 [-22.8 to 0.2]
  Percent change in TG at Week 48 (N=26) | -12.6 [-22.5 to -2.7]

12. Secondary Outcome: Percent Change in HDL-cholesterol (HDL-C) From Study Entry
Time Frame: Study entry and weeks 4, 12, 24, and 48
Population: All participants who initiated Atorvastatin and had HDL-C data available at study entry and the specified week.
Measure: Mean (90% Confidence Interval); unit: percentage of HDL-C at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 27
percentage of HDL-C at study entry
  Percent change in HDL-C at Week 4 (N=27) | 1.8 [-2.5 to 6.1]
  Percent change in HDL-C at Week 12 (N=27) | 2.3 [-1.1 to 5.7]
  Percent change in HDL-C at Week 24 (N=26) | 3.0 [-3.1 to 9.1]
  Percent change in HDL-C at Week 48 (N=26) | 4.2 [-3.5 to 11.9]

13. Secondary Outcome: Percent Change in Apolipoprotein A1 (Apo A-1) From Study Entry
Time Frame: Study entry and weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin and had Apo A-1 data available at study entry and the specified week.
Measure: Mean (90% Confidence Interval); unit: percentage of Apo A-1 at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 24
percentage of Apo A-1 at study entry
  Percent change in Apo A-1 at Week 12 (N=24) | 0.8 [-3.2 to 4.8]
  Percent change in Apo A-1 at Week 24 (N=23) | 2.4 [-2.7 to 7.5]
  Percent change in Apo A-1 at Week 48 (N=24) | 0.3 [-4.8 to 5.4]

14. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B) From Study Entry
Time Frame: Study entry and weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin and had Apo B data available at study entry and the specified week.
Measure: Mean (90% Confidence Interval); unit: percentage of Apo B at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 24
percentage of Apo B at study entry
  Percent change in Apo B at Week 12 (N=24) | -27.2 [-32.0 to -22.4]
  Percent change in Apo B at Week 24 (N=23) | -25.1 [-29.5 to -20.7]
  Percent change in Apo B at Week 48 (N=24) | -23.8 [-30.5 to -17.1]

15. Secondary Outcome: Percent Change in High-sensitivity CRP (Hs-CRP) From Study Entry
Time Frame: Study entry and weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin and had hs-CRP data available at study entry and the specified week.
Measure: Median (90% Confidence Interval); unit: percentage of hs-CRP at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 25
percentage of hs-CRP at study entry
  Percent change in hs-CRP at Week 12 (N=25) | 0 [-35 to 44]
  Percent change in hs-CRP at Week 24 (N=23) | -20 [-67 to 0]
  Percent change in hs-CRP at Week 48 (N=24) | 0 [-78 to 17]

16. Secondary Outcome: Percent Change in Interleukin 6 (IL-6) From Study Entry
Time Frame: Study entry and weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin and had IL-6 data available at study entry and the specified week.
Measure: Median (90% Confidence Interval); unit: percentage of IL-6 at study entry
Arm/Group | Atorvastatin
Number analyzed (Participants) | 24
percentage of IL-6 at study entry
  Percent change in IL-6 at Week 12 (N=24) | -1 [-32 to 110]
  Percent change in IL-6 at Week 24 (N=23) | -19 [-32 to -5]
  Percent change in IL-6 at Week 48 (N=24) | -11.5 [-34 to 46]

17. Secondary Outcome: Percentage of Participants With Undetectable Plasma HIV-1 RNA
Description: Undetectable is defined as plasma HIV-1 RNA below the lower limit of quantification of the assay used.
Time Frame: Study entry and weeks 12, 24, and 48
Population: All study participants who initiated Atorvastatin and had HIV-1 RNA data available at the specified week.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 28
percentage of participants
  Week 0 (N=28) | 71.0 [54.0 to 85.0]
  Week 12 (N=26) | 69.0 [51.0 to 84.0]
  Week 24 (N=26) | 62.0 [44.0 to 77.0]
  Week 48 (N=26) | 69.0 [51.0 to 84.0]

18. Primary Outcome: Percentage of Participants Experiencing at Least One Treatment-related Adverse Event (AE) by Age Group
Description: as for outcome 1
Time Frame: Study entry to weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 10 to 14 Years Old | 15 to 23 Years Old
Number analyzed (Participants) | 7 | 21
percentage of participants
  Week 12 | 14.3 [0.7 to 52.1] | 0 [0 to 13.3]
  Week 24 | 14.3 [0.7 to 52.1] | 0 [0 to 13.3]
  Week 48 | 28.6 [5.3 to 65.9] | 0 [0 to 13.3]

19. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE) by Age Group
Description: as for outcome 2
Time Frame: Study entry to weeks 12, 24, and 48
Population: All participants who initiated Atorvastatin.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 10 to 14 Years Old | 15 to 23 Years Old
Number analyzed (Participants) | 7 | 21
percentage of participants
  Week 12 | 14.3 [0.7 to 52.1] | 23.8 [9.9 to 43.7]
  Week 24 | 14.3 [0.7 to 52.1] | 23.8 [9.9 to 43.7]
  Week 48 | 28.6 [5.3 to 65.9] | 28.6 [13.2 to 48.7]

ADVERSE EVENTS:
Time Frame: From date of Atorvastatin initiation until Week 48.
Description: The DAIDS Adverse Event (AE) Grading Table (Version 1.0) was used for grading of AEs. Expedited adverse event reporting followed Version 2.0 of the DAIDS Expedited Adverse Event Manual.
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 3/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=28)
Pneumonia (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=28)
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Otorrhoea (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 4
Otitis media (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 11
Blood bilirubin increased (Investigations) | 6
Blood calcium increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 16
Blood glucose decreased (Investigations) | 6
Blood glucose increased (Investigations) | 2
Blood potassium decreased (Investigations) | 3
Blood sodium decreased (Investigations) | 5
Blood uric acid increased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 16
Neutrophil count decreased (Investigations) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Target enrollment was 40 participants (20 in each age cohort). However, the study was prematurely discontinued due to administrative reasons, having enrolled only 28 participants (21 participants aged 10 to 14 and 7 participants aged 15 to 23).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights